CLINICAL TRIAL: NCT04893395
Title: Assessment of the Impact of Clinical Pharmacogenomics on Real and Potential Medication Use in Veterans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Does not meet criteria for a clinical trial per IRB review.
Sponsor: Auburn University (Other)
Collaborators: Tuscaloosa Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Courtney Watts Alexander, Assistant Professor, Auburn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TVA_IRBNetID_1614352
Record Dates: First submitted 2021-05-12; First posted 2021-05-19 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Pharmacogenetics; Depressive Disorder, Major; Medication Therapy Management
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacogenomic Screening (Experimental): Eligible patients who verbally consent to participate will receive two pharmacogenomics telehealth visits.
  Interventions: Other: Pharmacogenomic Screening

INTERVENTIONS:
Other: Pharmacogenomic Screening — First telehealth appointment:
  1. Pharmacogenomics education and informed consent
  2. Medical history
  3. Sample collection
  Second telehealth appointment:
  1. Results of pharmacogenomic testing
  2. Utility and limitations of pharmacogenomic testing
  3. Patient-specific potential impacts on current or future medication therapies
  4. Answering of patient questions
  5. Referral to mental health provider(s) for treatment-specific recommendations

SUMMARY:
The purpose of this study is to assess the prevalence of veterans with major depressive disorder (MDD) who are being treated with a medication that has current Clinical Pharmacogenetics Implementation Consortium (CPIC) or Pharmacogenomics Knowledgebase (PharmGKB) actionable recommendations that have a pharmacogenomic variation that impacts the safety or efficacy of the subject medication.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years
2. Prescribed at least one chronic medication for mental health which is considered pharmacogenomically actionable, as defined above (amitriptyline, doxepin, imipramine, nortriptyline, citalopram, escitalopram, fluvoxamine, paroxetine, sertraline, or venlafaxine).
3. Diagnosis of major depressive disorder (MDD)

Exclusion Criteria:

1. Subject is a prisoner or is under a court order for treatment as part of a sentence or incarceration
2. Persistent medication non-adherence for reasons not potentially linked to pharmacogenomic variation (e.g. inability to obtain medications due to cost; non-adherence due to cognitive impairment)
3. Individuals receiving mental health treatment/care from a non-VA facility
4. Individuals who are terminally ill
5. Inability to communicate in and/or understand English

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of pharmacogenomic variation with actionable recommendations for medications currently utilized | At enrollment
  A medication history will be conducted at enrollment to ensure patient meets criteria for enrollment. Patients will provide a saliva sample at this timepoint. The rate of pharmacogenomic variation will be calculated based on current medications at enrollment; however, the pharmacogenomic screening panel may take up to 6 weeks to return to the patient and investigator.

SECONDARY OUTCOMES:
Rate of pharmacogenomic variation with actionable recommendations for all actionable medications | At enrollment
Mental health disease state control/progression utilizing disease state-specific validated tools | 3-, 6-, and 12-months post-recommendation via retrospective chart review
  Validated, disease state-specific tools will be utilized to assess control or progression. Specifically, depression control will be assessed utilizing PHQ-9 as documented within the chart. This will be assessed via retrospective chart review.
Medication-related costs | 3-, 6-, and 12-months post-recommendation via retrospective chart review
  Claims data will be used to assess medication-related costs at specific time points.
Medication-related adverse events | 3-, 6-, and 12-months post-recommendation via retrospective chart review
Number of primary care, mental health provider, mental health pharmacist, specialist, and emergency room visits and hospitalizations | 3-, 6-, and 12-months post-recommendation via retrospective chart review
Patient reported medication adherence and reasons for non-adherence | 3-, 6-, and 12-months post-recommendation via retrospective chart review
Patient reported reasons for non-adherence | 3-, 6-, and 12-months post-recommendation via retrospective chart review
Number of pharmacogenomic recommendations made and accepted | 3-, 6-, and 12-months post-recommendation via retrospective chart review
Type of pharmacogenomic recommendations made and accepted | 3-, 6-, and 12-months post-recommendation via retrospective chart review
Number of non-pharmacogenomic recommendations made and accepted | 3-, 6-, and 12-months post-recommendation via retrospective chart review
Type of non-pharmacogenomic recommendations made and accepted | 3-, 6-, and 12-months post-recommendation via retrospective chart review

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly B Lloyd, Pharm.D., Study Director — Auburn University
Locations (1):
- Tuscaloosa VAMC, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No